CLINICAL TRIAL: NCT06795776
Title: Efficacy and Safety of Eschscholzia Tablets in Adults with Insomnia Disorder Symptoms: a Monocentric, Randomized, Double-blind, Placebo-controlled, Parallel Group, Prospective Study
Brief Title: Eschscholzia Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: A. Vogel AG (Industry)
Collaborators: DCC Convex Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5'000'642
Record Dates: First submitted 2025-01-15; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Sleep

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum Group: Eschscholzia tablets (Experimental): One Escholzia tablet (1.0 g) contains as active pharmaceutical ingredient:
  0.503 g Eschscholzia californica Herba rec. tinct. conc. as the active pharmaceutical ingredient (API) corresponding 600 mg powdered herbal material.
  Interventions: Drug: Eschscholzia tablets
- Control Group: Placebo tablets (Placebo Comparator): A placebo tablet will be provided that matches the verum in its optical and sensorial properties and posology. Contains: microcrystalline cellulose, Colloidal anhydrous silica, glycerol distearate, caramel couleur and colorants.
  Interventions: Drug: Placebo Tablets

INTERVENTIONS:
Drug: Eschscholzia tablets — The intervention will be provided as swallowable "Eschscholzia tablets" (1.0 g) containing 0.503g Eschscholzia californica Herba rec. tinct. conc. as the active pharmaceutical ingredient (API) corresponding 600 mg powdered herbal material.
  Arms: Verum Group: Eschscholzia tablets
Drug: Placebo Tablets — A placebo tablet will be provided that matches the verum in its optical and sensorial properties and posology. Contains: microcrystalline cellulose, Colloidal anhydrous silica, glycerol distearate, caramel couleur and colorants.
  Arms: Control Group: Placebo tablets

SUMMARY:
This is a clinical study aimed at evaluating the efficacy and safety of Eschscholzia tablets in adults with insomnia disorder symptoms. The study will be conducted at one center, participants will randomly be assigned to either the treatment or placebo. Neither the participants, nor the researchers will know who is receiving the treatment (double-blind). The study is also placebo-controlled, meaning some participants receive a dummy pill instead of the actual treatment, and it involves a parallel-group design, where the treatment and placebo groups are studied at the same time. The study is exploratory, meaning it is investigating new possibilities and is not yet fully conclusive.

The purpose of this study is to determine main efficacy and safety of the newly developed herbal medicinal product Eschscholzia tablets. A total of 100 subjects will be enrolled in the study and assigned to either Eschscholzia tablets or placebo.

The Local Ethics Committee at the clinical site has given their approval for the study to be run.

Male or female participats aged between 18 and 75 years (inclusive), generally healthy and with a self reported history of disturbed sleep on at least 3 nights per week for at least the prior 1 month with a self-reported impact on daytime functioning are allowed to take part in the study.

Overall, the study has the following visits in the clinic, planned for each patient: Screening visit, Study centre Visit 2, Final study centre Visit 3. Between these visits participants will go through a "run-in" period (1 week between Visit 1 and 2) and treatment period (1 month between visit 1 and 3), both at home. Upon visit 2 participants will obtain the study product. They will be asked to administer a daily dose of 2 tablets (either Eschscholzia tablets or Placebo) over a 4-week period, starting from Visit 2 and continuing until Visit 3. Every intake of study product should be noted on the sleep diary pages that the participants obtain.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary, written, informed consent to participate in the study
* Self reported difficulty or maintaining sleep or waking too early, or daytime impairement or distress based on subject's information related to sleep pattern during at least the preceding month before screening.
* Self reported history of disturbed sleep on at least 3 nights per week for at least the last 1 month before screening.

  * ≥30 min to fall asleep
  * ≥30 min awake during sleep time
  * Self-reported total sleep time of ≤ 6.5 h
* ISI total score ≥ 10
* Confirmation of presence of insomnia diagnosis according to the ICD-10 F51.0/ICD-11 7A00 criteria by the physician upon anamnesis.
* Reported Impact on daytime functioning associated with sleep maintenance as measured with question 7 of the ISI, Score >= 2
* Freezing capacities available for storage of saliva samples.
* Willingness and infrastructure available to run aktigraphic device (bed sensor) properly

Exclusion Criteria:

* Body mass index (BMI) <18.0 or >30.0 kg/m2.
* Individual is pregnant, planning to be pregnant during the study period, lactating, or women of childbearing potential who are unwilling to commit to the use of a medically approved form of contraception throughout the study period.
* Any known acute organic disorder affecting sleep quality, such as narcolepsy, obstructive sleep apnea (OSA), restless leg syndrome (RLS), periodic limb movement syndrome (PLMS), circadian rhythm disorder, rapid-eye-movement behavior disorder, benign prostatic hyperplasia (BPH), urinary tract infections, irritated bladder, acute and/or chronic pain.
* Any known acute or chronic psychiatric condition (e.g., severe mono- or bipolar depression, history of suicidal ideation or attempt, severe anxiety disorders, severe personality disorders, borderline personality disorder, psychoses).
* Have a significant acute or chronic coexisting illness or any condition which contraindicates entry to the study in the opinion of the Investigator (e.g. migraines, active infections, renal insufficiency, hepatopathy, and dementia).
* History of alcohol or drug misuse
* Regular alcohol consumption exceeding 140g/week, heavy smoking (>10 cigarettes/day), high caffeine intake (>10 glasses/day).
* Current intake of drugs that could influence sleep (e.g., psychotropic, sedatives, hypnotics, nicotine-replacement therapies, over-the-counter sleep aids, hormone therapy, health products and oriental herbs (such as valerian, hops, passionflower, hypericum).
* Have a clinically significant high/low blood pressure (systolic over 159 mmHg, resp. lower than 80 mmHg or diastolic over 99 mmHg, resp. lower than 60 mmHg).
* History or planned travel to a different time zone within 1 month of the first visit or/and during the study participation.
* Shift-worker.
* Not fluent in local language.
* Have (known) hypersensitivity to plants from the poppy family (Papaveraceae) or known hypersensitivity to the active substance/s (Eschscholzia californica, microcrystalline cellulose, Colloidal anhydrous silica, sodium croscarmellose, glycerol distearate, caramel couleur and Ferrous(III) oxide).
* Participation in another study with any investigational product within 30 days of screening and during the intervention period.
* Investigator believes that the subject may be uncooperative and/or noncompliant and should therefore not participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Change between baseline and over 4-week treatment phase for perceived sleep quality as measured with the Insomnia Severity Index (ISI) | Change between baseline and over 4-week treatment phase
  Min: 0 score points, Max: 28 score points Lower scores mean better outcomes
Change in perceived sleep quantity/quality as per the daily sleep diary | Change between baseline and over 4-week treatment phase

SECONDARY OUTCOMES:
Change in physiological sleep quantity and quality as measured via actigraphy (bed sensor) | Change between baseline and over 4-week treatment phase
ISI Responder criteria assessed at the end of intervention on visit 3 | On Day 36
  ISI Responder criteria assessed at the end of intervention on visit 3 (day 36): a) Ratio of subjects with a ISI score reduction of ≥ 5 points from baseline, b) ratio of subjects achieving a ISI score reduction of at least 50% from baseline, c) Proportion of subjects reaching an ISI total score of ≤ 7, indicating no clinically significant insomnia symptoms, d) Proportion of subjects achieving the ISI composite score. ISI composite score criteria: the ISI composite score will be considered achieved if a subject meets at least two of the responder criteria a)-c); e) Ratio of subjects with an ISI score reduction of -8.4 or more score points
Change in daytime sleepiness symptoms severity as measured with the Epworth Sleepiness Scale (ESS) | Change between baseline and over 4-week treatment phase
  Min: 0 score points, Max: 24 score points Lower scores mean better outcomes
Change in Profile of Mood states as measured with the POMS-2 questionnaire (POMS-2) | Change between baseline and over 4-week treatment phase
  The POMS-2 includes the following primary scales:
  Tension-Anxiety Depression-Dejection Anger-Hostility Fatigue-Inertia Confusion-Bewilderment Vigor-Activity (positive scale)
  Higher raw scores on negative scales indicate greater mood disturbance. Higher raw scores on the Vigor-Activity scale indicate positive mood states.
Change in state anxiety as measured with the State-Trait-Anxiety-Inventory (STAI-Y1/Y2) | Change between baseline and over 4-week treatment phase
  STAI-Y1: Measures state anxiety (temporary and situational anxiety). STAI-Y2: Measures trait anxiety (general and long-standing anxiety tendencies).
  Both STAI-Y1 & STAI-Y2 are individually assessed as follows
  Minimum Score: 20 (low anxiety) Maximum Score: 80 (high anxiety)
  Lower scores mean better outcomes
Change in anxiety disorders as per the assessment of the clinician on the HAM-A scale (HAM-A) | Change between baseline and over 4-week treatment phase
  Minimum Score: 0 (no anxiety) Maximum Score: 56 (severe anxiety) Lower scores mean better outcomes
Change in psychological well-being as measured with the Depression, Anxiety, and Stress Scale (DASS-21). | Change between baseline and over 4-week treatment phase
  has 21 items, diivided into three subscales:
  Depression (7 items) Anxiety (7 items) Stress (7 items)
  Minimum Score per Subscale: 0 Maximum Score per Subscale (adjusted): 42
  lower scores mean better outcomes
Subjective efficacy | Day 36
  Patient's perceived efficacy will be assessed upon final visit 3 by asking the question how the subjects would rate the effectiveness of the study product to treat insomnia, sleeping problems and/or accompanying symptoms on a scale: "bad" = 0, "average" = 1, "good" = 2, "very good" = 3.
Subjective tolerability | On Day 36
  Patient's perceived tolerability will be assessed upon final visit 3 by asking the question how they rate their self-perceived tolerability of the IP on a scale: "bad" = 0, "average" = 1, "good" = 2, "very good" = 3.
Acceptance of the treatment | On day 36
  Patient's perceived acceptance is assessed upon final visit V3 by asking "would you take the test medication again to treat insomnia, sleeping problems and/or accompanying symptoms? Answers possible: "yes" or "no".
Rate/kind of adverse events | on day 36
Blood pressure | Change between baseline and day 36
  Blood pressure (BP):
  Systolic and diastolic BP will be assessed by using an automated BP measurement device.
Blood pulse | Change between baseline and day 36
  Blood pulse will be assessed by using an automated measurement device
Change in Blood safety parameters | Change between baseline and day 36
  The following factors will be analysed as per standard normal ranges for adults (f/m) by an external independent and certified medical diagnostic laboratory:
  * Red blood cell counts
  * Leukocytes counts /White blood cell count
  * Lymphocyte count
  * Thrombocyte count /Platelet counts
  * Monocyte count
  * Granulocyte count
  * Hemoglobin levels
  * Hematocrit levels
  * Mean corpuscular volume
  * Mean corpuscular hemoglobin
  * Mean corpuscular hemoglobin concentration
  * Glutamat-pyruvat-transaminase (GPT)
  * Glutamat-oxaloacetate-transaminase (GOT)
  * Gamma-glutamyltransferase (GGT)
  * Total bilirubin
  * Creatinine
  * Blood Glucose
  * Total Cholesterol
  * Erythrocyte sedimentation rate (ESR)
  * C-reactive protein (CRP)
Rate/kind of comedication | Change between baseline and day 36
Treatment compliance | on day 36
  Upon Visit 3, product intake compliance will be verified by counting the remaining tablets of the study product returned by subjects.
  Limits for subjects to be compliant is an intake of study product within 80% - 120% of the intended study product intake schedule.

CONTACTS AND LOCATIONS:
Locations (1):
- Diagnostics and Consultation Center Convex, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided
IPD may be sharaable upon reasonable request